CLINICAL TRIAL: NCT03932643
Title: A Phase 1 Trial of ONC-201 Maintenance Therapy in Acute Myeloid Leukemia and Myelodysplastic Syndrome After an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: ONC-201 Maintenance Therapy in Acute Myeloid Leukemia and Myelodysplastic Syndrome After Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0274-19-FB
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ONC-201 Treatment (Experimental): A 3+3 dose escalation design will be followed. Given the safety profile in prior trials, A dose of 250 mg weekly will be the starting dose. The first 12-15 patients are expected to receive escalating doses of ONC 201, the remaining patients will go on the expansion cohort.
  Interventions: Drug: ONC-201

INTERVENTIONS:
Drug: ONC-201 — ONC-201 Capsules, 125 mg
  Oral ONC-201 at various dose levels will be given at weekly intervals for up to 13 cycles (52 weeks); 4-week therapy will be considered 1 cycle.
  Other Names: dordaviprone

SUMMARY:
This is a single-center Phase 1 trial of 20 patients with AML/MDS. Eligible patients will be enrolled following an informed consent between 6-20 weeks after allogeneic hematopoietic stem cell transplant. Patients will receive weekly oral ONC 201 for a total of 52 weeks.

DETAILED DESCRIPTION:
This is a single-center Phase 1 trial of 20 participants with AML/MDS. Eligible participants will be enrolled following an informed consent between 6-20 weeks after allogeneic hematopoietic stem cell transplant. Participants will receive weekly oral ONC-201 for a total of 52 weeks.

The objectives of the study are: 1. To determine the safety and preliminary efficacy of ONC-201 maintenance therapy among partcipants with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS), who undergo allogeneic hematopoietic stem cell transplant.

Participants will be monitored for toxicities (using Common Terminology Criteria for Adverse Events, CTCAE version 5.0), quality of life [Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT)], and immunologic changes. We will also examine changes in functional status (Karnofsky Performance Scale (KPS), instrumental activities of daily living and short physical performance battery), rates of disease relapse and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. A history of Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) with at least one of the following features:

   AML: High-risk AML as defined by the 2017 European LeukemiaNet criteria (e.g. complex karyotype with ≥3 changes), AML with high-risk mutations (e.g. TP53, RUNX1, or ASXL1 mutations), transplant being performed in second remission or beyond, or AML with active disease or minimal residual disease positivity before or after transplant.

   MDS: MDS with high or very-high risk cytogenetic changes as defined by the Revised International Prognostic Scoring System (e.g. complex karyotype with ≥3 changes),53 the presence of TP53 mutation, high-risk or very high-risk MDS not responding to 4 cycles of hypomethylating agents, MDS progressing following initial response, persistence of MDS after transplant, or transplant being performed in second remission or beyond.
2. Receipt of allogeneic hematopoietic stem cell transplant 6-20 weeks prior to enrollment
3. Disease status: <5% bone marrow blast at the time of enrollment
4. All donor sources and conditioning regimens are allowed
5. Adults, Age ≥19 years (for the state of Nebraska)
6. Karnofsky Performance Status (KPS) of ≥70
7. Absolute neutrophil count (ANC) greater than 1000/µL without the use of granulocyte colony stimulating factor in the past 2 weeks, and platelet count 50,000/µL without platelet transfusion in the past 2 weeks.
8. Able to take oral medication.
9. Female patient of reproductive potential must have a negative serum or urine pregnancy test ≤7 days prior to starting the study drug.
10. Male and female patients of reproductive potential must be willing to avoid pregnancy or fathering children from enrollment to two months after the end of study treatment. This will require either a total abstinence, OR exclusively non-heterosexual activity (when this is in line with the preferred and usual lifestyle of the subject), OR two methods of contraception
11. Written informed consent to participate in the study.

Exclusion Criteria:

1. A history of acute graft-versus-host disease grade III/IV or initiation of any new immunosuppressive agent for treatment of graft-versus-host disease within 4 weeks prior to enrollment. Oral beclomethasone or budesonide, empirically used for possible but not biopsy-proven graft-versus-host disease, will not be considered an exclusion criterion.
2. Use of prednisone at a dose of ≥0.25 mg/kg/day (or equivalent dose of another glucocorticoid) at the time of enrollment
3. Active uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection
4. Presence of known HIV infection, active hepatitis B or C infection.
5. Total bilirubin, aspartate transaminase, alanine transaminase 2 X the upper limit of the normal range. Patients with elevated bilirubin secondary to Gilbert syndrome will not be excluded.
6. Creatinine clearance <30 mL/min
7. Presence of uncontrolled cardiopulmonary conditions such as ongoing cardiac arrhythmias, unstable angina or myocardial infarction, New York Heart Association class III/IV congestive heart failure, or severe chronic obstructive pulmonary disease or other pulmonary condition resulting in a requirement of supplemental oxygen or having a resting O2 saturation <90% by pulse oximetry
8. Pregnancy or breastfeeding.
9. Known hypersensitivity, or intolerance to any of the study medications, or excipients.
10. Treatment with any other investigational agent, device, or procedure, within 21 days (or 5 half-lives, whichever is greater)
11. Patients on dopamine antagonists for treatment of psychotic disorder or Parkinson's disease will be excluded. A brief use of drugs such as clozapine or haloperidol for a few days for treatment of nausea or other indication will not be prohibited. The use of tricyclic antidepressants does not constitute an exclusion criterion.
12. Any other condition that is judged by the physician to potentially interfere with compliance to the study protocol or pose a significant risk to the patient.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities during the first cycle | after one month of treatment
  The rate of dose limiting toxicities during the first cycle (among the dose escalating cohort)
Grade ≥3 toxicities | during the first 3 cycles ot treatment (each cycle is 28 days)
  The number of grade ≥3 toxicities

SECONDARY OUTCOMES:
Number of toxicities (all grades) during the duration of maintenance therapy with ONC 201 | upto 13 months after initiation of ONC 201
  Number of toxicities (all grades) associated with the use of ONC 201 during the entire duration of maintenance therapy with ONC 201
The rate of relapse | upto 2 years after enrollment
  The rate of relapse
The rate of relapse-free survival | upto 2 years after enrollment
  The rate of relapse-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya R Bhatt, MBBS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No